CLINICAL TRIAL: NCT01115153
Title: Prophylaxis With Single Versus Five Dose of Antibiotic Therapy as Treatment of Patients With Gangrenous Acute Appendicitis (Randomized, Controlled Clinical Trial)
Brief Title: Prophylaxis With Single Versus Five Dose of Antibiotic Therapy as Treatment of Patients With Gangrenous Acute Appendicitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Industrial de Santander (Other)
Collaborators: Hospital Universitario de Santander (Unknown)
Responsible Party: Principal Investigator, Henry Uscategui Cristancho, General Surgeon, Universidad Industrial de Santander
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 74186942
Record Dates: First submitted 2010-04-19; First posted 2010-05-04 (Estimated); Last update posted 2011-08-23 (Estimated); Status verified 2011-08

CONDITIONS: Gangrenous Appendicitis
Keywords: Acute appendicitis; Antibiotic prophylaxis; Wound infection; Nosocomial infection
MeSH Terms: conditions — Appendicitis; Wound Infection; Cross Infection | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Antibiotic prophylaxis (Experimental): Rate of Wound infection in patients with gangrenous appendicitis with single doses of antibiotic (before surgery)
  Interventions: Other: prophylaxis
- Antibiotic treatment, wound infection (Active Comparator): Rate of Wound infection in patients with gangrenous appendicitis with five days antibiotic therapy (after surgery)
  Interventions: Other: therapy

INTERVENTIONS:
Other: prophylaxis — single doses of antibiotics before surgery in patients with gangrenous appendicitis Metronidazole 500 mg IV + amikacin 1 gr IV
  Arms: Antibiotic prophylaxis
Other: therapy — antibiotic treatment (5 days) therapy in patients with gangrenous appendicitis metronidazole 500 mg IV three times a day + amikacin 1 gr IV per day
  Arms: Antibiotic treatment, wound infection

SUMMARY:
A prospective, randomized controlled clinical trial was conducted at the Hospital Universitario de Santander to test the effectiveness of providing a single 1-dose therapy of antibiotic prophylaxis versus a 5-day antibiotic therapy in patients with acute gangrenous appendicitis.

DETAILED DESCRIPTION:
Introduction: For patients with acute gangrenous appendicitis, it is common to provide antibiotics during 5-7 days in order to reduce the incidence of infection of the surgical wound; however the benefit of such treatment has not been tested. A prospective, randomized controlled clinical trial was conducted at the Hospital Universitario de Santander to test the effectiveness of providing a single 1-dose therapy of antibiotic prophylaxis versus a 5-day antibiotic therapy in patients with acute gangrenous appendicitis.

Materials and Methods: From December 2007 to November 2009, 799 patients went through surgery after being diagnosed with acute appendicitis. Out of this set, 150 patients diagnosed with acute gangrenous appendicitis, were randomly assigned to one of two groups: control group (group A: 72 patients received a 5-day antibiotic therapy), and treatment group (group B: 78 patients received a single 1-dose of antibiotic prophylaxis). The experimental outcomes included: the incidence of infection of the surgical wound, the length of the hospital stay, and the adverse effects derived from a prolonged use of antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* patients with diagnosis of acute appendicitis with intraoperative finding of a gangrenous appendix who accepted to enter the study

Exclusion Criteria:

* patients under 12 or older 65 years old
* Patients with possible immunosuppression such as diabetes, cancer, kidney failure, liver failure
* Pregnancy
* Patients who have received antibiotic treatment within seven days before surgery
* Patients difficult to monitor or follow up

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2007-12; Primary Completion 2009-11 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
wound infection | 30 days
  Signs of surgical wound infection as heat, pain, erythema and secretion with involvement of skin,subcutaneous tissue and organ or space

SECONDARY OUTCOMES:
Length of the hospital stay | 30 days
  Duration in days from admission until discharge
Adverse effects treatment related | 30 days
  Adverse effects derived from the usage of antibiotics

CONTACTS AND LOCATIONS:
Overall Officials: Henry A Uscategui, Physician, Principal Investigator — Universidad Industrial de Santander; Francisco Camacho, Physician, Study Director — Universidad Industrial de Santander
Locations (1):
- Hospital Universitario de Santander, Bucaramanga, Santander Department, Colombia

REFERENCES:
- [Background] Ein SH, Sandler A. Wound infection prophylaxis in pediatric acute appendicitis: a 26-year prospective study. J Pediatr Surg. 2006 Mar;41(3):538-41. doi: 10.1016/j.jpedsurg.2005.11.052. PMID 16516631
- [Background] Gollin G, Abarbanell A, Moores D. Oral antibiotics in the management of perforated appendicitis in children. Am Surg. 2002 Dec;68(12):1072-4. PMID 12516811
- [Background] Bauer T, Vennits B, Holm B, Hahn-Pedersen J, Lysen D, Galatius H, Kristensen ES, Graversen P, Wilhelmsen F, Skjoldborg H, et al. Antibiotic prophylaxis in acute nonperforated appendicitis. The Danish Multicenter Study Group III. Ann Surg. 1989 Mar;209(3):307-11. doi: 10.1097/00000658-198903000-00010. PMID 2647050
- [Result] Rucinski J, Fabian T, Panagopoulos G, Schein M, Wise L. Gangrenous and perforated appendicitis: a meta-analytic study of 2532 patients indicates that the incision should be closed primarily. Surgery. 2000 Feb;127(2):136-41. doi: 10.1067/msy.2000.101151. PMID 10686977
- [Result] Lemieur TP, Rodriguez JL, Jacobs DM, Bennett ME, West MA. Wound management in perforated appendicitis. Am Surg. 1999 May;65(5):439-43. PMID 10231213
- [Result] Taylor E, Berjis A, Bosch T, Hoehne F, Ozaeta M. The efficacy of postoperative oral antibiotics in appendicitis: a randomized prospective double-blinded study. Am Surg. 2004 Oct;70(10):858-62. PMID 15529837
- [Result] Page CP, Bohnen JM, Fletcher JR, McManus AT, Solomkin JS, Wittmann DH. Antimicrobial prophylaxis for surgical wounds. Guidelines for clinical care. Arch Surg. 1993 Jan;128(1):79-88. doi: 10.1001/archsurg.1993.01420130087014. PMID 8418785
- [Result] Gorecki WJ, Grochowski JA. Are antibiotics necessary in nonperforated appendicitis in children? A double blind randomized controlled trial. Med Sci Monit. 2001 Mar-Apr;7(2):289-92. PMID 11257737
- [Result] Andersen BR, Kallehave FL, Andersen HK. Antibiotics versus placebo for prevention of postoperative infection after appendicectomy. Cochrane Database Syst Rev. 2005 Jul 20;2005(3):CD001439. doi: 10.1002/14651858.CD001439.pub2. PMID 16034862
- [Result] Mui LM, Ng CS, Wong SK, Lam YH, Fung TM, Fok KL, Chung SS, Ng EK. Optimum duration of prophylactic antibiotics in acute non-perforated appendicitis. ANZ J Surg. 2005 Jun;75(6):425-8. doi: 10.1111/j.1445-2197.2005.03397.x. PMID 15943731
- [Result] Snelling CM, Poenaru D, Drover JW. Minimum postoperative antibiotic duration in advanced appendicitis in children: a review. Pediatr Surg Int. 2004 Dec;20(11-12):838-45. doi: 10.1007/s00383-004-1280-x. Epub 2004 Oct 6. PMID 15480707
- [Result] Gleisner AL, Argenta R, Pimentel M, Simon TK, Jungblut CF, Petteffi L, de Souza RM, Sauerssig M, Kruel CD, Machado AR. Infective complications according to duration of antibiotic treatment in acute abdomen. Int J Infect Dis. 2004 May;8(3):155-62. doi: 10.1016/j.ijid.2003.06.003. PMID 15109590
- [Result] Hoelzer DJ, Zabel DD, Zern JT. Determining duration of antibiotic use in children with complicated appendicitis. Pediatr Infect Dis J. 1999 Nov;18(11):979-82. doi: 10.1097/00006454-199911000-00009. PMID 10571434
- [Result] Almqvist P, Leandoer L, Tornqvist A. Timing of antibiotic treatment in non-perforated gangrenous appendicitis. Eur J Surg. 1995 Jun;161(6):431-3. PMID 7548380